CLINICAL TRIAL: NCT02870621
Title: Volume of Perirenal Fat and Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 12-PP-06
Record Dates: First submitted 2016-07-29; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The perirenal fat may alter renal function by secreting fibrotic inflammatory agents when accumulates during obesity. Nephrectomy for renal tumor is a model that would provide tissue samples to test this hypothesis. Renal tumor could itself be responsible for inflammation and fibrosis in its environment. This study aims to measure the influence of the tumor on his kidney Environment and fat and define molecular markers not influenced by renal tumor. The main objective is to compare the inflammation of the perirenal fat taken in two locations in the same patient, in contact and 4 cm from the outer edge of the tumor, each patient as his own control. The secondary objective is to compare the degree of interstitial fibrosis of the renal cortex in the same sampling methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Indication nephrectomy for kidney tumor
* Stadium T1a, T1b or T2 and M0 according to the TNM (Tumor Nodes Metastasis) classification of tumors

Exclusion Criteria:

* Nephrectomy indication for chronic pyelonephritis
* Asian topic because of the difference threshold values used to characterize the metabolic syndrome in this population
* Diabetes type I or II due to a high score of renal interstitial fibrosis
* Infection with HIV (Human immunodeficiency virus)
* Partial nephrectomy (a part of the kidney on the side of the tumor is left in place)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment is in hospital, all patients being hospitalized in case of nephrectomy for kidney cancer. The treatment will be done like habitually and fat will be sample.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Numbers of renal interstitial fibrosis | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No